CLINICAL TRIAL: NCT02922816
Title: A Pilot Study Using Fecal Microbiota Transplant in Renal Transplant Recipients to Eliminate Multidrug-Resistant Organism Colonization After Infection and Examine Gastrointestinal Carriage in a Randomized Placebo-Controlled Design
Brief Title: FMT for MDRO Colonization After Infection in Renal Transplant Recipients
Acronym: PREMIX
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was paused and was not resumed due to the COVID-19 pandemic.
Sponsor: Emory University (Other)
Collaborators: Cepheid (Industry)
Responsible Party: Principal Investigator, Colleen S. Kraft, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00090101
Record Dates: First submitted 2016-09-27; First posted 2016-10-04 (Estimated); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Infection Due to Resistant Organism
Keywords: Carbapenem-resistant Enterobacteriaceae (CRE); Vancomycin-resistant Enterococcus (VRE); Multidrug Resistant Organism (MDRO); Fecal Microbiota Transplant (FMT); Renal Transplant; Colonization; Infection; Antibiotic Resistance; Resistome; Multidrug Resistant (MDR) Pseudomonas
MeSH Terms: conditions — Infections; Pseudomonas Infections | interventions — Fecal Microbiota Transplantation; Cathartics; Defecation; Angptl4 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control arm (Placebo Comparator): The control arm will participate in the bowel preparation and stool or perirectal swab sampling but will not receive Fecal Microbiota Transplant (FMT) nor will they be fasting during their first study cycle (Cycle 0). Participants testing positive for a multi-drug resistant organism at the of Cycle 0 will be eligible to receive microbiota restoration transplant (MRT) for up to two cycles, as necessary (Cycles 1 and 2).
  Interventions: Procedure: Bowel preparation; Procedure: Stool or perirectal swab sampling
- Fecal Microbiota Transplant (FMT) (Experimental): The experimental arm will participate in the bowel preparation, stool or perirectal swab sampling, and will receive Fecal Microbiota Transplant (FMT) using Allogeneic Human Stool in Glycerol 10% (AHSG) on Day 1 of each cycle (Cycles 1 and 2).
  Interventions: Biological: Fecal Microbiota Transplant (FMT); Procedure: Bowel preparation; Procedure: Stool or perirectal swab sampling; Other: Fasting

INTERVENTIONS:
Biological: Fecal Microbiota Transplant (FMT) — The Fecal Microbiota Transplant (FMT) using Allogeneic human stool in glycerol (10%) (AHSG) intervention will be administered via rectal retention enema and performed in either an inpatient or outpatient clinic.
  Arms: Fecal Microbiota Transplant (FMT)
Procedure: Bowel preparation — Trial participants will undergo the bowel preparation by taking magnesium citrate the day before the cycle begins (Day -1).
Procedure: Stool or perirectal swab sampling — Stool or perirectal swabs will be collected at screening (for eligibility determination) and Days 1, 2, 15, and 36 of each cycle.
Other: Fasting — In Cycle 1 and Cycle 2, participants cannot consume food, alcohol, or other liquids on Day 1 prior to the intervention. Trial participants will not be fasting on Day 1 of Cycle 0.
  Arms: Fecal Microbiota Transplant (FMT)

SUMMARY:
Transplant patients are at increased risk of colonization and infection with Multidrug Resistant Organisms (MDROs) due to medications that modify their immune systems, increased healthcare and antibiotic exposure, and surgical manipulation of mucosa. In this study, kidney transplant patients who have infections with resistant bacteria will be given a Fecal Microbiota Transplant (FMT), also known as a fecal transplant, after they receive antibiotic treatment. This study will see if FMT will eliminate the resistant bacteria so that the kidney transplant patients do not have to use last resort antibiotics.

This Phase 1 pilot study is to obtain preliminary safety data for FMT in renal transplant patients to support the rationale for a subsequent clinical trial, not to establish efficacy or toxicity. This trial is designed to test the safety of FMT, identify clinical outcomes, assess feasibility, and refine the target population in participants with MDRO colonization and intestinal dysbiosis. Data from this study should provide directions for the design of future clinical trials.

DETAILED DESCRIPTION:
Potential participants who meet key eligibility criteria [adults who have undergone renal transplantation and have a history of infection with the Target Multidrug Resistant Organisms (MDRO)] will be approached for consideration of study participation. For this study, Target MDRO colonization is defined as a positive bacterial culture of either carbapenem-resistant Enterobacteriaceae (CRE), vancomycin-resistant Enterococcus (VRE), Extended Spectrum Beta-Lactamases (ESBL), and/or multidrug resistant (MDR) Pseudomonas from stool or perirectal swab sampling.

The 20 trial participants will be randomized in a 1:1 ratio to one of two arms: the control arm [not receiving Allogeneic Human Stool in Glycerol (10%; AHSG) via Fecal Microbiota Transplant (FMT)] and the experimental arm (receiving AHSG via FMT). Participants in the control arm participants can crossover to receive the treatment after completing a study cycle without FMT. Each cycle lasts 6 weeks and participants will complete a maximum of 2 treatment cycles; participants randomized to the experimental arm will complete a maximum of two cycles and those randomized to the control arm will complete up to three cycles. Upon completion of the final cycle, all trial participants will be followed for just over 6 months.

In addition to the trial participants, there will also be one stool donor participant. The consented, screened, and eligible stool donor will be identified from an established group of stool donors and will undergo screening procedures that are specific to this study. This individual will donate human stool for the preparation of the AHSG (known as the investigational new drug (IND) product for this study). Upon processing of AHSG, the stool donor will enter the Follow-Up Period and remain available for communication to the study team (if necessary) until the Study Completion Date. However, no scheduled study assessments are required of the stool donor.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign a written informed consent document.
* Ability and willingness to comply with study protocol requirements and receive an enema.
* History of MDRO infection with at least one of the following target MDROs: CRE, VRE, ESBL, or MDR Pseudomonas.
* Prior receipt of a renal transplant.
* If applicable, willingness to discontinue probiotics or other microbiota restoration therapies during screening at least seven days prior to study Day 1.
* The effects of FMT on the developing human fetus are unknown. For this reason, women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* Negative blood or urine human chorionic gonadotropin (hCG) testing on the day of FMT for WOCBP with documentation of negative test result.
* Negative baseline Human Immunodeficiency Virus (HIV) test.
* Known serology CMV status confirmed by Medical History (if positive). If no mention of positivity in medical records, serology is tested within 30 days of enrollment for:

  * Cytomegalovirus (CMV) by polymerase chain reaction (PCR)
  * Cytomegalovirus (CMV), serology Immunoglobulin G (IgG)

Exclusion Criteria:

* Female participants who are pregnant, breastfeeding, lactating, or planning a pregnancy during study duration (through 4 weeks after the last dose of investigational product).
* Prior gastrointestinal surgery or intervention:

  * Ileostomy (in the last 3 months)
  * Colostomy (in the last 3 months)
  * Gastric or colon resection (in the last 3 months)
  * Bariatric surgery (any prior history)
  * Total colectomy (any prior history)
* Any of the following gastrointestinal conditions:

  * Irritable Bowel Syndrome (IBS) with diarrhea in the last 12 months
  * Crohn's disease
  * Ulcerative Colitis
  * Celiac disease
  * Untreated in-situ colorectal cancer
  * Microscopic colitis
  * Toxic megacolon or ileus
  * Tube feeding (current or planned)
* Known positive stool studies or cultures in the last 30 days for: Ova or parasites, Salmonella, Shigella, Campylobacter
* Other enteropathogens - defined as any positive result other than C. difficile on the Biofire FilmArray gastrointestinal panel, (Campylobacter, Plesiomonas, Salmonella, Vibrio, Yersinia, Enteroaggregative Escherichia coli (EAEC), Enteropathogenic Escherichia coli (EPEC), Enterotoxigenic Escherichia coli (ETEC), Shigella, Cryptosporidium, Cyclospora, Entamoeba, Giardia, Adenovirus, Astrovirus, Norovirus, Rotavirus, Sapovirus).
* Known uncontrolled intercurrent illness(es) such as, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Acute coronary syndrome
  * Cardiac arrhythmia
* Any other intercurrent acute illness that in the opinion of the investigator will preclude subject from entering the study
* On systemic antibiotics for any reason other than recent MDRO infection. If a potential participant is taking antibiotics for treatment (not prophylaxis) of MDRO infection, then the participant must complete the planned antibiotic course by study Day -2.
* Compromised immune system other than transplant immunosuppression:

  * HIV-positive as identified by one of the following: Positive HIV test, prior diagnosis of HIV, or active or history of administration of antiretroviral therapy (ART) other than for pre-exposure prophylaxis or post-exposure prophylaxis.
  * Known Absolute Neutrophil (ANC) <1000 neutrophils per cubic millimeter (mm^3) in the last 3 months
  * Active malignancy requiring intensive induction chemotherapy, radiotherapy, or biologic treatment either concurrently or in the last 2 months
  * Acute leukemia
  * History of hematopoietic cell transplantation, either allogeneic or autologous in the last 3 years
* History of solid organ transplant rejection in the last 6 months
* Significant food allergy to foods that are part of the stool donor participant's diet.
* Life expectancy is 24 weeks or less.
* Any condition that, in the opinion of the investigator, might interfere with study objectives or limit compliance with study requirements, including but not limited to:

  * Known active intravenous drug or alcohol abuse
  * Psychiatric illness
  * Social situation
* Participated in an investigational study that also meets one of the following criteria:

  * Received an interventional agent (drug, device, or procedure) in the last 28 days
  * Enrollment on this study or any other interventional study for MDROs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | Up to 30 weeks
  The safety and feasibility of using FMT in adult participants with Target MDRO colonization after infection will be measured by comparing the number of adverse events (assessed by CTCAE v4.0) after Day 1 of each cycle as compared to baseline.
Change in Target MDRO Growth | Day 1, Up to 30 weeks
  The primary outcome is target MDRO growth on perirectal swab or stool culture on Day 36 of each cycle compared Screening and Day 1 culture results. Participants will be classified as having a complete response, partial response, refractory response or progression based on their Day 36 culture results. Partial response, refractory response, and progression may be collapsed in a non-response category for analytic purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen S Kraft, MD, MSc, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified sequencing data may be made available to outside collaborators upon request and approval by study team.
Access Criteria: Researchers interested in using data collected in this study should submit a methodologically sound protocol to the study PI.

REFERENCES:
- [Result] Woodworth MH, Conrad RE, Haldopoulos M, Pouch SM, Babiker A, Mehta AK, Sitchenko KL, Wang CH, Strudwick A, Ingersoll JM, Philippe C, Lohsen S, Kocaman K, Lindner BG, Hatt JK, Jones RM, Miller C, Neish AS, Friedman-Moraco R, Karadkhele G, Liu KH, Jones DP, Mehta CC, Ziegler TR, Weiss DS, Larsen CP, Konstantinidis KT, Kraft CS. Fecal microbiota transplantation promotes reduction of antimicrobial resistance by strain replacement. Sci Transl Med. 2023 Nov;15(720):eabo2750. doi: 10.1126/scitranslmed.abo2750. Epub 2023 Nov 1. PMID 37910603
- [Derived] Woodworth MH, Kwon JH, Kraft CS. An Ounce of Prevention Is Equivalent to How Much Decolonization Exactly? Clin Infect Dis. 2021 Jun 1;72(11):e924. doi: 10.1093/cid/ciaa1524. No abstract available. PMID 33029623